CLINICAL TRIAL: NCT04498520
Title: Phase I Trial of Abexinostat Combined With Palbociclib and Fulvestrant in Patients With Antiestrogen Refractory ER+, HER2- Breast Cancer and Gynecological Metastatic Tumors
Brief Title: Abexinostat, Palbociclib, and Fulvestrant for the Treatment of Breast or Gynecologic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Pamela Munster (Other)
Collaborators: Pfizer (Industry); Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pamela Munster, Prinicpal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20953; NCI-2020-05026 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Hormone Receptor Positive Breast Carcinoma; Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Metastatic Endometrioid Adenocarcinoma; Metastatic Fallopian Tube Carcinoma; Metastatic HER2 Negative Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Ovarian Carcinoma; Metastatic Primary Peritoneal Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Refractory Breast Carcinoma; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8
Keywords: Metastatic Breast Cancer; Gynecological Cancer; HER2 Negative; Antiestrogen Refractory ER+
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Endometrioid; Fallopian Tube Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms | interventions — Fulvestrant; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (abexinostat tosylate, palbociclib, fulvestrant) (Experimental): Patients receive abexinostat PO BID on days 1-4, 8-11, and 15-18, palbociclib PO QD on days 1-21, and fulvestrant IM on days 1 and 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abexinostat Tosylate; Drug: Fulvestrant; Drug: Palbociclib

INTERVENTIONS:
Drug: Abexinostat Tosylate — Given PO
  Other Names: PCI-24781 Tosylate
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991

SUMMARY:
This phase I trial investigates the side effects and best dose of abexinostat and palbociclib when given together with fulvestrant in treating patients with breast or gynecologic cancer. Abexinostat may prevent tumor cells from growing and multiplying and may kill tumor cells. Palbociclib may prevent or slow the growth of tumor cells when used with other anti-hormonal therapy. Estrogen can cause the growth of breast and gynecologic tumor cells. Fulvestrant may help fight breast or gynecologic cancer by blocking the use of estrogen by the tumor cells. Giving abexinostat, palbociclib, and fulvestrant may work better in treating patients with breast or gynecologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To determine the safety and tolerability of abexinostat tosylate (abexinostat) and palbociclib in combination with fulvestrant.
2. To determine the maximum tolerated dose (MTD) for abexinostat and palbociclib when combined with fulvestrant at standard dose.

SECONDARY OBJECTIVES:

1. To describe the pharmacokinetics associated with abexinostat.
2. To describe the efficacy of abexinostat and palbociclib in combination with fulvestrant in patients with antiestrogen refractory estrogen receptor positive (ER+), HER2 negative(-) breast cancer and gynecological metastatic tumors.
3. To assess the clinical benefit rate (CBR) defined as complete response (CR), partial response (PR), and stable disease (SD) at 6 months and progression free survival according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

EXPLORATORY OBJECTIVES:

1. To assess correlations between overall response rate (ORR), CBR at 6 months, and progression free survival (PFS) with genomic aberrations assessed as cell free tumor deoxyribonucleic acid (DNA) and histone acetylation on peripheral blood.
2. To assess correlations between ORR, CBR at 6 months, and PFS endpoints and peripheral blood mononuclear cell (PBMC) histone deacetylase (HDAC) gene expression, PBMC acetylation in vivo and ex vivo.

OUTLINE: This is a dose-escalation study of abexinostat and palbociclib.

Patients receive abexinostat orally (PO) twice daily (BID) on days 1-4, 8-11, and 15-18, palbociclib PO once daily (QD) on days 1-21, and fulvestrant intramuscularly (IM) on days 1 and 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients will be followed for 90 days after completion of treatment or removal from study, or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* BREAST CANCER: Participants must have histologically confirmed hormone receptor (HR)+, HER2- locally advanced or metastatic stage IV breast cancer. HER2- should be defined as 0 or 1 by immunohistochemistry, or HER2 gene amplification by fluorescence in situ hybridization (FISH), chromogenic in situ hybridization (CISH), or in situ hybridization (ISH) performed upon the primary tumor or metastatic lesion (ration < 2 and HER2 copy < 4). Estrogen receptor (ER) and progesterone receptor (PR) expression positivity is defined as more than 5% of tumor cells nuclei positive by immunohistochemistry in the sample on testing
* BREAST CANCER: Patients must have had disease progression after treatment with anti-estrogen therapy combined with Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor after a minimum of at least 3 months therapy in the metastatic setting and no more than 3 prior lines of systemic therapy for metastatic breast cancer (MBC), unrestricted prior therapy in the dose escalation

  * Note: Patients with breast cancer who were not previously treated with CDK4/6 inhibitors or have not tolerated full doses of prior ribociclib or palbociclib or abemaciclib are not eligible
* ENDOMETRIAL CANCER: Patients must have histologically confirmed metastatic endometrial cancer of endometrioid type
* ENDOMETRIAL CANCER: Tumors must have ER expression
* ENDOMETRIAL CANCER: Patients must have received a maximum of one line of hormonal therapy for the treatment of endometrial cancer and may have received any lines of chemotherapy treatment

  * Note: Mixed tumor histology is allowed if the non-endometrioid component is less than 1%. Tumor must be estrogen receptor positive
* OVARIAN, FALLOPIAN TUBE, OR PERITONEAL EPITHELIAL CANCER: Patients must have histologically confirmed recurrent or metastatic ovarian, fallopian, or peritoneal epithelial carcinoma
* OVARIAN, FALLOPIAN TUBE, OR PERITONEAL EPITHELIAL CANCER: Tumors must have ER expression
* OVARIAN, FALLOPIAN TUBE, OR PERITONEAL EPITHELIAL CANCER: Patients must have received a maximum of one line of hormonal therapy for the treatment of ovarian cancer and may have received any lines of chemotherapy treatment

  * Note: pure clear cell and pure mucinous ovarian carcinomas are not eligible
* ALL PATIENTS
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1
* Leukocytes >= 2,500/microliter (mcL)
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin > 9 g/dl (transfusions are allowed if more than 7 days prior to enrollment)
* Platelets >= 100,000/mcL
* Total bilirubin < upper limit of normal (ULN) except for patients with Gilbert's syndrome, who may only be included if the total bilirubin is =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN
* International normalized ratio (INR) =< 1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug)
* Aspartate transaminase (AST) < 2.5 x ULN, except for patients with liver metastasis, who are only included if the AST is < 5 x ULN
* Alanine transaminase (ALT) < 2.5 x ULN, except for patients with liver metastasis, who are only included if the ALT is < 5 x ULN
* Alkaline phosphate =< 2.5 x ULN (unless bone metastasis is present in the absence of liver metastasis, in which 3.0 x ULN would be acceptable)
* Serum creatinine =< 1.5 mg/dl
* Patients must be recovered from the effects of any prior surgery, radiotherapy, or other antineoplastic therapy
* Patients may have received fulvestrant if the duration of response was more than 3 months
* Ability to understand a written informed consent document, and the willingness to sign it
* All female patients must be post-menopausal or rendered postmenopausal during the therapy
* All male patients must be surgically sterile or agree to abstain from sperm donation and use both, a highly effective contraception with child bearing potential female partners (implants, injectables, combined oral contraceptives, some intrauterine device (IUD)s, sexual abstinence) and a barrier method (e.g., condoms, cervical rings, cervical condoms, sponge) during participation in the study and for 90 days after the last dose of study drug
* Must be able to swallow pills

Exclusion Criteria:

* Patient with symptomatic visceral disease or any disease burden that renders the patient ineligible for endocrine therapy per the investigator's best judgment
* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse event to grade 1 or less from agents administered more than 2 weeks earlier
* Patient has received treatment with any investigational drug within 21 days prior to study treatment administration. For classes of investigational agents that are not known to have prolonged toxicities, the washout time may be decreased to 14 days at the discretion of the principal investigator
* Patients may not have any known intolerability to any of the involved agents or established cytopenias to CDK4/6 inhibitors that require dose modifications or dose delays of greater than 2 weeks
* Patient with a known hypersensitivity to any of the excipients of palbociclib, abexinostat, or fulvestrant, including to peanut and soy
* Patient has a concurrent malignancy or malignancy within 3 years of study entry, with the exception of adequately treated, basal or squamous cell skin carcinoma, nonmelanomatous skin cancer or curatively resected cervical cancer
* Patient who has a history of untreated brain, or leptomeningeal, metastases (central nervous system (CNS) imaging is not required before study entry unless there is a clinical suspicion of CNS involvement)
* Participants with previously treated brain metastases may participate, provided:

  * They are stable (without evidence of progression by imaging for at least four weeks and any neurologic symptoms have returned to baseline)
  * They have no evidence of new or enlarging brain metastases (confirmed by imaging within 28 days of the first dose of study drug)
  * They are not using steroids for at least 7 days before the first dose of study drug
  * Have isolated lesions that were treated with localized radiation therapy

    * This exception does not include leptomeningeal metastases, which is excluded regardless of clinical stability
* Patient must not have been previously treated with histone deacetylase inhibitor (HDACi), with the exception of low dose of divalproex sodium (Depakote) or valproic acid
* Patient has any medical, psychiatric or social condition, which in the opinion of the investigator, places the patient at an unacceptably high risk for toxicities or affects compliance to study procedures
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient is currently receiving or has received systemic therapeutic doses of corticosteroids =< 2 weeks prior to starting study drug, or has not fully recovered from side effects of such treatment

  * Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patient has known clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Patient is currently receiving any of the following substances and cannot be discontinued 30 days prior to cycle 1 day 1:

  * Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pummelos, star fruit, Seville oranges) and their juices that are strong inducers or inhibitors of CYP3A4/5,
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5 and CYP2D6 substrates
* Has uncontrolled intercurrent illness including, but not limited to:

  * Uncontrolled infection
  * Disseminated intravascular coagulation
  * Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | At the end of Cycle 1 (each cycle is 28 days)
  An occurrence of any of the protocol specified toxicities occurring during cycle 1: (1) Hematologic - Grade 4 neutropenia lasting > 5 consecutive days, Grade 3/4 febrile neutropenia, Grade 4 thrombocytopenia lasting >=7 days, or Grade 3 or 4 thrombocytopenia w/ clinically significant bleeding or requirement for platelet transfusion, (2) Non-hematologic: Any adverse event (AE) >= Grade 3, with the exceptions of Grade 3 nausea, vomiting, diarrhea, clinically insignificant laboratory abnormality, or fatigue resolving to Grade <=2 w/in 72 hours (3) Any AE that results in delay in administration of abexinostat or palbociclib of less than 75% and a delay of more than 7 days before starting cycle 2 unless the AE can be clearly attributed to an extraneous cause. DLTs are classified according to Medical Dictionary for Regulatory Activities (MedDRA) version 20 and graded for severity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE).
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 28 days)
  Defined as the dose at which fewer than one-third of participants experience a DLT or the highest dose at which no more than one instance of DLT is observed among 6 participants treated.
Incidence of treatment-related adverse events (AE) | From initiation of study treatment until 30 days after completion of study treatment, up to 1 year
  Adverse events will be classified using MedDRA version 20.0 and graded for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Abexinostat: Maximum concentration (Cmax) | Cycle 1, Days 1 and 11; Cycle 2, Day 11 (each cycle is 28 days)
  Serum samples will be collected in order to obtain the Cmax of abexinostat over the course of 2 cycles under the following schedule: Pre-dose, immediately post-admin, 4 hrs (+/- 30 min) post-start of drug administration, and after completion of study drug administration on Cycle 1, Day 11 and Cycle 2, Day 11
Abexinostat: Trough concentration (Ctrough) | Cycle 1, Days 1 and 11; Cycle 2, Day 11 (each cycle is 28 days)
  Serum samples will be collected in order to obtain the Ctrough of abexinostat over the course of 2 cycles under the following schedule: Pre-dose, immediately post-admin, 4 hrs (+/- 30 min) post-start of drug administration, and after completion of study drug administration on Cycle 1, Day 11 and Cycle 2, Day 11
Objective response rates (ORR) | Up to 1 year
  An objective response is defined as Complete Response (CR), Partial Response (PR), assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 from initiation of study therapy until disease progression or study discontinuation, . ORR will be estimated using an exact method based on the binomial distribution (Clopper-Pearson interval) with a 90% confidence interval.
Clinical benefit rate (CBR) | Up to 6 months
  CBR is defined as the proportion of participants who displayed a clinical benefit (CR, PR, or Stable Disease (SD)) per RECIST v 1.1 and without disease progression at 6 months after initiation of study therapy.
Median progression-free survival (PFS) | Up to 1 year
  PFS will be determined according to RECIST v 1.1 and measured as the time from first objective response after initiation of study therapy until the time of progression or death, which ever occurs first . Will be estimated using Kaplan-Meier analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela N Munster, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No